CLINICAL TRIAL: NCT01073449
Title: Action Elicited By Scheduled In-Hospital Follow-Up of Cardiac Devices
Brief Title: Actions Elicited by In-hospital Follow-up of Cardiac Devices
Acronym: ATHENS
Status: Completed | Type: Observational
Sponsor: Cliniche Humanitas Gavazzeni (Other)
Responsible Party: U.O. Aritmologia - Cliniche Humanitas Gavazzeni, Dr. Giosuè Mascioli
Other Study IDs: GAVBS1
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Results first posted 2011-02-28 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-01

CONDITIONS: Cardiac Pacemaker, Artificial; Implantable Cardioverter-Defibrillator
Keywords: Cardiac devices; In-Hospital Follow-up; Analytical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac device: All patients implanted with a cardiac device, pacemaker(PM)or Implantable Cardioverter Defibrillator (ICD)
  Interventions: Procedure: In-hospital follow-up of cardiac device

INTERVENTIONS:
Procedure: In-hospital follow-up of cardiac device — Electrical measures taken during normal follow-up and clinical status of the patient

SUMMARY:
This study will enroll all patients who will attend an in-hospital follow-up of cardiac device since February 22nd 2010 to June 21st 2010.

Primary objective of the study is to observe how many of patients seen during these period (approximately 5000) will receive a change in cardiac device programming or in drug therapy or a scheduled or urgent hospital admission.

These data should help to clarify how useful and safe is a remote monitoring strategy for this kind of patients.

DETAILED DESCRIPTION:
Number of Pacemakers (PM) and Implantable Cardioverter Defibrillators (ICD) is rapidly growing due to enlarged indications. This fact causes an exponential increase in scheduled in-hospital follow-ups. For this reason, all the companies that produce PM and ICD have released systems that allow remote monitoring and follow-up of cardiac devices (both PM and ICD) and U.S. guidelines have already been changed, in order to suggest remote follow-up of these devices at appropriated intervals.

Nevertheless, informations on actions taken during scheduled in-hospital follow-up are incomplete.

ATHENS study has been designed to answer to 3 questions:

1. How often, during a scheduled in hospital follow-up physicians "change" something ? (device programming; drug therapy; scheduled device replacement ...)
2. The "rate of change" is different is the follow-up is required pby the general practitioner who normally takes care of the patients or by the patient itself?
3. Change are more frequent during PM or during ICD follow-up or during cardiac resynchronization therapy devices?

ELIGIBILITY:
Inclusion Criteria:

* All patients with a cardiac device

Exclusion Criteria:

* Follow-up of a cardiac device at discharge from hospital after first implant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who will undergo an in-hospital follow-up of a cardiac device
Sampling Method: Probability Sample
Enrollment: 3362 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giosue Mascioli, MD, Study Chair — Cliniche Humanitas Gavazzeni; Antonio Curnis, MD, Study Chair — Spedali Civili di Brescia; Maurizio Landolina, MD, Principal Investigator — Policlinico San Matteo Pavia; Gian-Paolo Gelmini, MD, Principal Investigator — Ospedale Civile di Desenzano d/Garda; Franco Ruffa, MD, Principal Investigator — Ospedale A. Manzoni - Lecco
Locations (8):
- Italy (8):
  - U.O. Aritmologia - Cliniche Humanitas Gavazzeni, Bergamo, Bergamo
  - Laboratorio di Elettrofisiologia - Spedali Civili, Brescia, Brescia
  - Laboratorio di Elettrofisiologia, Desenzano del Garda, Brescia
  - Laboratorio di Cardiologia - Ospedale Civile, Casalmaggiore, Cremona
  - Laboratorio di Elettrofisiologia - Ospedale A. Manzoni, Lecco, Lecco
  - Laboratorio di Elettrofisiologia, Merate, Lecco
  - Laboratorio di Elettrofisiologia - Ospedale Carlo Poma, Mantova, Mantova
  - Laboratorio di Elettrofisiologia - Ospedale San Matteo, Pavia, Pavia

REFERENCES:
- [Background] Senges-Becker JC, Klostermann M, Becker R, Bauer A, Siegler KE, Katus HA, Schoels W. What is the "optimal" follow-up schedule for ICD patients? Europace. 2005 Jul;7(4):319-26. doi: 10.1016/j.eupc.2005.02.117. PMID 15944090
- [Background] Fauchier L, Sadoul N, Kouakam C, Briand F, Chauvin M, Babuty D, Clementy J. Potential cost savings by telemedicine-assisted long-term care of implantable cardioverter defibrillator recipients. Pacing Clin Electrophysiol. 2005 Jan;28 Suppl 1:S255-9. doi: 10.1111/j.1540-8159.2005.00071.x. PMID 15683509
- [Result] Brugada P. What evidence do we have to replace in-hospital implantable cardioverter defibrillator follow-up? Clin Res Cardiol. 2006;95 Suppl 3:III3-9. doi: 10.1007/s00392-006-1302-x. PMID 16598602
- [Derived] Mascioli G, Curnis A, Landolina M, Klersy C, Gelmini GP, Ruffa F; ATHENS Investigators. Actions elicited during scheduled and unscheduled in-hospital follow-up of cardiac devices: results of the ATHENS multicentre registry. Europace. 2011 Dec;13(12):1766-73. doi: 10.1093/europace/eur233. Epub 2011 Jul 14. PMID 21764815

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac Device: All patients implanted with a cardiac device (PM or ICD)
Period: Overall Study
Arm/Group | Cardiac Device
Started | 3362
Completed | 3362
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Device
Number analyzed (Participants) | 3362
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 640
  >=65 years | 2718
Age Continuous [Mean (Standard Deviation); unit: years] | 73.36 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1156
  Male | 2206
Region of Enrollment [Number; unit: participants]
  Italy | 3362

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients -Amongst Those Implanted With a Pacemaker - in Whom Something (Therapy, Device Programming ...) Has Been Changed During In-hospital Follow-up
Time Frame: 4 months
Population: 2246 represents the number of patients in the whole population that were implanted with a PM
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cardiac Device
Number analyzed (Participants) | 2246
Participants | 512 [492 to 532]

2. Primary Outcome: Number of Patients of the Whole Population in Whom Something (Therapy, Device Programming ...) Has Been Changed During In-hospital Follow-up
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cardiac Device
Number analyzed (Participants) | 3362
Participants | 767 [719 to 816]

3. Secondary Outcome: Number of Patients - Amongst Those Implanted With an Implantable Cardioverter Defibrillator (ICD)- in Whom Something (Therapy, Device Programming ...) Has Been Changed During In-hospital Follow-up
Time Frame: 4 months
Population: 693 represents the number of patients implanted with an ICD within the whole population
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cardiac Device
Number analyzed (Participants) | 693
Participants | 129 [128 to 130]

ADVERSE EVENTS:
Arm/Group | Cardiac Device
Serious Adverse Events (participants affected / at risk) | 0/3362
Other Adverse Events (participants affected / at risk) | 0/3362

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No